CLINICAL TRIAL: NCT00409123
Title: Effect of Systemic Cooling in Vasospasms (Kühleffekte Beim Vasospastischen Syndrom)
Brief Title: Effect of Systemic Cooling in Vasospasms
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Selim Orguel, MD, University Hospital, Basel, Switzerland
Other Study IDs: 007-KRK-2004-001
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Vasospastic Syndrome
Keywords: vasospastic women; controls; core cooling; core warming; external cooling; external warming; LDF; choroidal blood flow; temperature; vasospastic subjects; normal subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study tests whether women with Vasospastic Syndrome (VS) react more intensive than controls with distal vasomotions and choroidal blood flow changes to internal cooling/warming and external cooling/warming.

DETAILED DESCRIPTION:
Distal vasomotions and choroidal blood flow changes to internal cooling/warming and external cooling/warming was studied in VS and controls.Core cooling was induced by drinking of 250g ice/water mixture (4°C). Core warming was induced by drinking of 250g warm water (55°C). The study was controlled with respect to posture and room temperature.

ELIGIBILITY:
Inclusion Criteria:

* women
* luteal phase or contraceptives
* 19-35 years

Exclusion Criteria:

* somatic diseases
* psychiatric diseases
* BMI > 25
* BMI < 18

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: vasospastic women
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
LDF blood flow | repeated after each challenge
LDF velocity | repeated after each challenge
finger skin temperature | repeated after each challenge
core body temperature | repeated after each challenge
corneal temperature | repeated after each challenge

SECONDARY OUTCOMES:
subjective sleepiness | repeated after each challenge
subjective ratings of thermal comfort | repeated after each challenge

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orguel, MD, Study Director — Unversity Eye Clinic Basel
Locations (1):
- University Eye Clinic, Basel, Basel, Switzerland